CLINICAL TRIAL: NCT03508856
Title: Clinical and Histologic Evaluation of Picato 0.15% Gel in the Cosmetic Improvement of Photoaged Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skin Laser & Surgery Specialists (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, David J. Goldberg, MD, MD, Skin Laser & Surgery Specialists
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENC_008776
Record Dates: First submitted 2016-05-26; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Actinic Keratosis; Photo-aged Skin
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Gels

ARMS (1):
- Picato 0.015% gel (Experimental): Picato 0.015% gel, is a topical treatment for actinic ketatoses.
  Interventions: Drug: Ingenol Mebutate (Picato®) 0.015% gel

INTERVENTIONS:
Drug: Ingenol Mebutate (Picato®) 0.015% gel

SUMMARY:
Clinical Evaluation:

Subjects having actinic keratoses and meeting Glogau Photoaging Class III or IV complete the FDA approved 3 day course of Picato® 0.015% gel as approved for the treatment of facial Actinic Keratosis. Each subject undergoes clinical multiple-angle standardized photographs on day 1, day 7, day 30, and day 60. Full face photography will be obtained with the medical research digital camera. Both subjects and investigators complete questionnaires at each visit with individual questions regarding improvement in actinic keratoses and overall skin appearance, wrinkling, dyschromia, erythema, and textural quality of skin. Each characteristic listed above will be graded on a 5 point scale ranging from 0 (lowest quality/worst appearance) to 5 (highest quality/best appearance). In addition, investigators will examine the subject's face and assign a numeric assessment on a 9 point scale ranging from 0 to 8 using previously published verified Griffiths' Photonumeric Photoaging scale. A second and third investigator will be presented at random blinded pretreatment (day 0) and posttreatment (day 60) photographs of each subject and be asked to assign a numerical value from Griffiths' Photonumeric Photoaging Scale. These blinded investgators will be given no information regarding which day each photograph represents. Comparison will be made of skin quality questionnaire scores from each visit and the pre and post treatment Griffiths' Photonumeric Grades.

The investigator opted against a split-face study design given the difficulty of blinding with this type of study as well as difficulty recruiting subjects willing to treat for two separate courses.

Histologic Evaluation:

Standard 3mm dermatology punch biopsies from clinically sun damaged skin will be taken. Biopsy will be taken from either the cosmetically acceptable pre-or infra-auricular area. A digital photograph will be taken and used to identify the pre-treatment biopsy site. Biopsies will be taken of 5 subjects before treatment and at day 60. Day 60 biopsies will be taken immediately adjacent to previously photographed and identified pre-treatment biopsies. Biopsies will be stained with hematoxylin and eosin and histologic features of pre and post treatment skin will be evaluated. Measurement of actinic keratoses, solar elastosis and overall epidermal and dermal thickness pre and post treatment will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adults aged 45-75 years of age.
* Subjects must be in good general health as confirmed by the medical history.
* Subjects must be able to read, sign, and understand the informed consent.
* Subjects must meet the criteris for Glogau Photoaging class III or class IV.
* Subjects have a diagnosis of actinic keratosis.
* Subjects must be willing to apply Picato 0.015% gel
* Subjects must be willing to forego any other treatments on the face, including cosmetic treatments, tanning bed use, and excessive sun exposure while enrolled in the study.
* If a subject is a female of childbearing potential she must have a urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.

Exclusion Criteria:

-. Subjects with a history of melanoma anywhere on the body.

* Subjects with any unstable medical condition as determined by the clinical investigator.
* Subjects with untreated non-melanoma skin cancer on the face or within the treatment area.
* Subjects with dermatitis or any dermatologic disease in the treatment area that would obscure the evaluation of photoaging parameters.
* Subjects who have undergone any form of 'field treatment' including 5-fluorouracil, photodynamic therapy, or ingenol mebutate in the preceeding six months.
* Women who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects who have experienced a major medical event (including stroke, heart attack, etc) within 90 days of starting the study.
* Subjects who have active substance abuse disorders.
* Subjects who have known allergies to any components of the study drug.
* Subjects who are currently particpating in another clinical trial or who have completed a study involving laser, systemic, or topical treatment of the face within 30 days prior to study treatment initiation.
* Subjects who have received any of the following within 90 days prior to study treatment initiation:
* Interferon or interferon inducers
* Cytotoxic drugs
* Immunomodulators or immunosuppressive treatments (except inhaled or intranasal corticosteroids)
* Oral or parenteral corticosteroids
* Topical steroids to treatment area
* Any dermatologic procedures or surgeries to the treatment area, including cryosurgery for AKs
* Subjects who have used any topical prescription medications on the study area within 30 days prior to study treatment initiation

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2016-08-09 (Actual); Study Completion 2016-08-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the improvement in actinic keratoses and photoaged skin as measured numerically by Griffiths' Photonumeric Photoaging scale and questionnaires, | 60 days